CLINICAL TRIAL: NCT04420364
Title: Maintenance Versus Reduction of Immunosuppression for Renal Transplant Patients Hospitalized With COVID-19 Disease
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Decline in COVID cases
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Finnian McCausland, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020P001516
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: COVID; Kidney Transplant; Complications; Immunosuppression
MeSH Terms: interventions — Maintenance

STUDY DESIGN:
Intervention Model Description: Single-blind, parallel-group, randomized, active-controlled trial
Who Masked: Outcomes Assessor
Masking Description: This is a single-blind trial, in that only the assessor will be blinded to the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maintenance of Immunosuppression (Experimental): Maintenance of immunosuppression (defined as no change to pre-admission immunosuppression, or reduction in anti-metabolite by up to 50% (to a minimum of MMF 500 mg per day or azathioprine 50 mg per day)
  Interventions: Other: Maintenance or reduction of immunosuppression
- Reduction of Immunosuppression (Active Comparator): Reduction of immunosuppression (defined as anti-metabolite withdrawal plus reduction of tacrolimus or cyclosporin, to a minimum target trough concentration of 3 ng/mL for tacrolimus and 50 ng/mL for cyclosporin).
  Interventions: Other: Maintenance or reduction of immunosuppression

INTERVENTIONS:
Other: Maintenance or reduction of immunosuppression — Maintenance versus reduction of immunosuppression

SUMMARY:
This will be a randomized trial of maintenance versus reduction in immunosuppression in adult patients (age >18 years old) with functioning renal transplants admitted to hospital with confirmed COVID-19 disease.

DETAILED DESCRIPTION:
The optimal management of immunosuppression in renal transplant patients with COVID-19 disease is unclear. On one hand, many centers advocate reduction of immunosuppression in infected patients, with the rationale that such an approach will unleash the anti-viral T-cell response. However, on the other hand, some centers advocate there may be rationale to maintain baseline immunosuppression in order to mitigate against development of an uncontrolled over-activation of the immune response. The investigators propose to address this knowledge gap by performing a randomized clinical trial that will test formal comparisons of maintenance versus reduction in immunosuppression.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years
* COVID positive by RT-PCR or serology
* ≥ 6 months post-transplant
* use of anti-metabolite (mycophenolate or azathioprine) and calcineurin inhibitor (cyclosporin or tacrolimus)
* informed consent; first admission during study period
* participation within 72 hours of hospitalization

Exclusion Criteria:

* ICU care or need for invasive ventilation or use of pressors at screening/randomization
* COVID-19 disease severity score more than 5 at screening/randomization
* Known donor specific antibody
* eGFR <20ml/min/1.73m2
* hematocrit <24%
* biopsy proven and treated rejection within last 3 months
* institutionalized individuals (prisoners)
* pregnancy
* participation in another clinical study with an investigational medicinal product within 30 days or within 5 half-lives of such, whichever is longer, prior to randomization and during the study
* any other conditions, which, in the opinion of the investigator would make the subject unsuitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Change in IL-6 concentration from baseline to day 7 | baseline to day 7

SECONDARY OUTCOMES:
Change in IL-6 concentration from baseline to day 28 | Baseline to day 28
Change in T cell response to SARS-CoV-2 | Baseline to day 7 and day 28
Change in titer of serum anti-SARS-CoV-2 antibodies | Baseline to day 7 and day 28
Change in COVID-19 disease severity score (range 1 to 8; higher worse) | Through day 28
Proportion of patients needing non-invasive ventilation or intubation | Through day 28
Proportion of patients developing ANC < 500 cells per microliter | Through day 28
Proportion of patients developing lymphopenia < 400 cells per microliter | Through day 28
Length of hospital stay | Through day 28
Proportion of patients developing biopsy-proven acute rejection | Through day 28
In-hospital and 28-day mortality | Through day 28
Adverse and serious adverse events | Through day 28

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Azzi, MD, PhD, Principal Investigator — Birgham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No